CLINICAL TRIAL: NCT01713127
Title: Efficacy and Safety of Remifentanil in Preterm Infants Who Require Ventilator Support
Brief Title: Remifentanil in Ventilated Preterm Infants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: declined enrollment
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); DongGuk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RFTN-02; 12077 (Other: Korea FDA)
Record Dates: First submitted 2012-08-31; First posted 2012-10-24 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2012-10

CONDITIONS: Preterm Infants; Mechanical Ventilator Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 5% dextrose infusion for 72 hours during ventilator care start within 48 hours after birth
  Interventions: Drug: Placebo
- remifentanil (Active Comparator): 0.1mcg/kg/min remifentanil infusion for 72 hours during ventilator care start within 48 hours after birth
  Interventions: Drug: remifentanil infusion

INTERVENTIONS:
Drug: remifentanil infusion
  Arms: remifentanil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of remifentanil in preterm infants during ventilator care with remifentanil and to analyze pharmacokinetics in preterm infants

ELIGIBILITY:
Inclusion Criteria:

* preterm infants (<37weeks of gestational age)
* requiring ventilator care
* informed consent

Exclusion Criteria:

* major anomaly
* 48hrs after birth
* requiring operation during drug infusion
* cord blood pH < 7.0
* intraventricular hemorrhage grade III or more
* investigators decision

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
premature infant pain profile (PIPP) | 24hours after remifentanil/placebo infusion
  PIPP measure during tracheal suction window period ; +/- 1hr

SECONDARY OUTCOMES:
intraventricular hemorrhage | up to 1 week of age
  intraventricular hemorrhage documented by sonography
pneumothorax | up to 1 week of age
  pneumothorax documented by X-ray or sonography
bronchopulmonary dysplasia | 28 days of age
  O2 dependency
duration of ventilator care | up to 4 months of age
  mechanical ventilator dependency
hospital day | upto 4 months of age
  days from admission to discharge from neonatal intensive care unit
time to full feeding | up to 2 months of age
  day of life when the baby reaches full enteral feeding, defined as a volume above 120 mL/kg/day
mortality | up to 4 months of age
  in-hospital death
development of adverse effects | from the start of remifentanil infusion to 1 hour after end of infusion
  category of adverse effects
  1. General appearance Fever or Hypothermia, Rash
  2. Respiratory & Cardiovascular Arrhythmia Tachypnea (RR >100/min) Desaturation (SpO2 <80%) Hypotension (inotropics use or need volume challenge) Bradycardia (HR <80/min) Tachycardia (HR >200/min)
  3. Gastrointestinal Abdominal distension Bilious gastric remain Vomiting Bloody Stool Necrotizing Enterocolitis
  4. Renal Oliguria (U/O < 1.0cc/kg/day)
  5. Neurologic Seizure Cerebral infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea